CLINICAL TRIAL: NCT01732653
Title: V-TIME: A Treadmill Training Program Augmented by Virtual Reality to Decrease Fall Risk in Older Adults, Patients With Parkinson's Disease and Individuals With Mild Cognitive Impairments
Brief Title: A Treadmill Training Program Augmented by Virtual Reality to Decrease Fall Risk in Older Adults
Acronym: VTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Newcastle University (Other); University Medical Center Nijmegen (Other); Universita degli Studi di Genova (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-12-NG-0505-CTIL; VTIME
Record Dates: First submitted 2012-11-05; First posted 2012-11-26 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Elderly Adults; Parkinson; Mild Cognitive Disorder
Keywords: virtual reality,; falls,; elderly,; Parkinson's disease,; MCI
MeSH Terms: conditions — Neurocognitive Disorders; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TT+VR (Experimental): The training will consist of walking on the treadmill while negotiating obstacles in a virtual reality simulation.Training will be provided3 times a week for a duration of 6 weeks (total of 18 sessions).
  Interventions: Other: TT+VR
- TT alone (Active Comparator): The training will consist of walking on the treadmill 3 times a week for a duration of 6 weeks (total of 18 sessions).
  Interventions: Other: TT alone

INTERVENTIONS:
Other: TT+VR — subjects will be walking on a treadmill while negotiating virtual obstacles provided by a computer simulation. The virtual environment will consist of obstacles, different pathways, narrow corridors and distracters, requiring modulations of step amplitude in two planes (i.e., height and width) coordinated with walking behaviour. The speed, orientation, size, frequency of appearance and shape of the targets will be manipulated according to individual needs following a standardized protocol.
  Other Names: training on a treadmill with virtual reality
  Arms: TT+VR
Other: TT alone — The participants will walk on the treadmill, their gait speed over-ground will be measured at the beginning of each week of training. Progression will include increasing the duration of each of the walking bouts and increasing walking speed.
  Other Names: treadmill training
  Arms: TT alone

SUMMARY:
The proposed randomized controlled trial will evaluate the effects of treadmill training augmented with virtual reality on fall risk.

300 older adults with a history of falls will be recruited to participate in this study. This will include older adults (n=100), patients with mild cognitive impairment (MCI) (n=100), and patients with Parkinson's disease (PD)(n=100). Subjects will be randomly assigned to the intervention group (treadmill training with virtual reality) or to the active-control group (treadmill training without virtual reality). Each person will participate in a training program set in an outpatient setting 3 times per week for 6 weeks. Assessments will take place before, after, and 1 month and 6 months after the completion of the training.

DETAILED DESCRIPTION:
A prospective, single blinded, parallel group, randomized controlled trial with 6 month follow-up will be employed to investigate the effects of treadmill training augmented with virtual reality on fall risk. The study will include 300 older participants who have experienced two or more falls in the previous 6 months. Participants will be randomized to either the intervention or control group. The intervention group will receive 18 sessions of Treadmill Training with Virtual Reality (TT+VR) and the active control comparison will receive 18 training sessions of treadmill training alone (TT) without the VR simulation All interventions will be delivered by therapists trained in the standard protocols. All subjects will be trained 3 times a week for 6 weeks, each session will last approximately 45 minutes.Training progression will be based on increasing both motor and cognitive challenges, individualized to the participant's level of performance.

Primary outcome measures:

The primary outcome measure of the study is fall rate for 6 months post intervention. Secondary outcome measures will include gait speed and gait variability under usual and dual task conditions and while negotiating physical obstacles will be measured. Endurance will be assessed using the 2 Minute Walk Test and mobility will be assessed using the Four Square Step Test (FSST), The Short Physical Performance Battery (SPPB) and the mini-Balance Evaluation Systems Test (mini-BESTest). Community ambulation will be assessed using a tri-axial accelerometer ('Axivity' Ltd.)which will be worn by the participants for 7 days. Cognitive function will be assessed using a computerized neuropsychological test battery (Mindstreams, 'NeuroTrax' Corp., NJ) as well as standardized neuropsychological tests (Montreal Cognitive Assessment,The Trail Making Test; Verbal Fluency). Quality of life will be evaluated using the SF-36 Health Survey

ELIGIBILITY:
Inclusion Criteria:

* 2 or more falls within 6 months prior to the beginning of the study
* Aged 60-85 years
* Able to walk for 5 minutes unassisted
* Adequate hearing and vision capabilities.
* Stable medication for the past 1 month and anticipated over a period of 6 months

Exclusion Criteria:

* Psychiatric co-morbidity
* Clinical diagnosis of dementia or other severe cognitive impairment (MMSE<24)
* History of stroke, traumatic brain injury or other neurological disorders (other than PD and MCI, for those groups)
* Acute lower back or lower extremity pain, peripheral neuropathy, rheumatic and orthopaedic diseases
* Unstable medical condition in the past 6 months
* Unable to comply with the training
* Interfering therapy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Falls rate | 6 months post intervention
  The primary outcome measure of the study is fall rate. Participants will keep a falls calendar for 6 months post intervention. Each time the participant falls he/she will tick the date on the calendar. These calendars will be returned to the researchers once a month in a pre-addressed envelope.

SECONDARY OUTCOMES:
Gait | 6 months post intervention
  Gait speed and gait variability under usual and dual task conditions and while negotiating physical obstacles will be measured. Participants will be asked to walk in a well-lit corridor under 3 conditions each of 1 minute: i) walking in a comfortable speed, ii) walking while subtracting 3s from a predefined number (dual task), iii) walking while negotiating two obstacles placed on the floor at specific locations. Spatial-temporal gait characteristics (e.g., gait speed (m/s), stride length (m), stride time (s), swing time (%), asymmetry, and step width (cm)) will be determined. Endurance will be assessed using the 2 Minute Walk Test.
Cognitive function | 6 months post intervention
  Cognitive function will be assessed using a computerized neuropsychological test battery (Mindstreams, NeuroTrax Corp., NJ). In addition, we will also include standardized neuropsychological tests such as the Montreal Cognitive Assessment (MoCA); The Trail Making Test (TMT) and the Verbal Fluency test.
Balance and mobility | 6 months post intervention
  The Four Square Step Test (FSST), The Short Physical Performance Battery (SPPB) and the mini-Balance Evaluation Systems Test (mini-BESTest) will be used to assess mobility. Community ambulation will be assessed using The Physical Activity Scale for the Elderly (PASE) and a tri-axial accelerometer (Axivity Ltd.) which will be worn by the participants for 7 days to quantify and monitor stepping and physical activity.
Quality of life | 6 months post intervention
  The SF-36 Health Survey, a generic self-report questionnaire designed to address health related quality of life will be used. Fear of Falling will be evaluated using the Falls Efficacy Scale-International.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Hausdorff, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (5):
- Department of Rehabilitation Sciences, Katholieke Universiteit Leuven, Leuven, Belgium
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Department of Neurosciences Universita Degli Studi Di Genova, Italy, Genova, Italy
- Department of Geriatric Medicine and Neurology, Radboud University Nijmegen Medical Center The Netherlands, Nijmegen, Netherlands
- Institute for Aging and Health, University of Newcastle, UK, Newcastle, United Kingdom

REFERENCES:
- [Derived] Maidan I, Hacham R, Galperin I, Giladi N, Holtzer R, Hausdorff JM, Mirelman A. Neural Variability in the Prefrontal Cortex as a Reflection of Neural Flexibility and Stability in Patients With Parkinson Disease. Neurology. 2022 Feb 22;98(8):e839-e847. doi: 10.1212/WNL.0000000000013217. Epub 2021 Dec 14. PMID 34906983
- [Derived] Droby A, Maidan I, Jacob Y, Giladi N, Hausdorff JM, Mirelman A. Distinct Effects of Motor Training on Resting-State Functional Networks of the Brain in Parkinson's Disease. Neurorehabil Neural Repair. 2020 Sep;34(9):795-803. doi: 10.1177/1545968320940985. Epub 2020 Jul 18. PMID 32684069
- [Derived] Mirelman A, Rochester L, Maidan I, Del Din S, Alcock L, Nieuwhof F, Rikkert MO, Bloem BR, Pelosin E, Avanzino L, Abbruzzese G, Dockx K, Bekkers E, Giladi N, Nieuwboer A, Hausdorff JM. Addition of a non-immersive virtual reality component to treadmill training to reduce fall risk in older adults (V-TIME): a randomised controlled trial. Lancet. 2016 Sep 17;388(10050):1170-82. doi: 10.1016/S0140-6736(16)31325-3. Epub 2016 Aug 11. PMID 27524393
- [Derived] Mirelman A, Rochester L, Reelick M, Nieuwhof F, Pelosin E, Abbruzzese G, Dockx K, Nieuwboer A, Hausdorff JM. V-TIME: a treadmill training program augmented by virtual reality to decrease fall risk in older adults: study design of a randomized controlled trial. BMC Neurol. 2013 Feb 6;13:15. doi: 10.1186/1471-2377-13-15. PMID 23388087